CLINICAL TRIAL: NCT07294716
Title: VITAL - "Visual Improvement With Toric Asymmetrical Lenses": Enhancing Vision in Irregular Corneas
Brief Title: Improving Visual Quality in Patients With Irregular Corneas Using Asymmetrical Toric Intraocular Lenses
Acronym: VITAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUK-Ophthalmology-017
Record Dates: First submitted 2025-12-01; First posted 2025-12-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Irregular Astigmatism; Astigmatism; Cataract and IOL Surgery
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMILens Individual Implantation (Active Comparator): An acrylic hydrophilic, one piece 4-loop haptic, monofocal, toric IOL (AMILens Individual, AMIPLANT GmbH, Germany) will be implanted into the capsular bag after removal of the of the natural lens. This IOL is CE-certified. Asphericity and dioptric power of the IOL are customized for each individual eye.
  Interventions: Device: AMILens Individual

INTERVENTIONS:
Device: AMILens Individual — An acrylic hydrophilic, one piece 4-loop haptic, monofocal, toric IOL (AMILens Individual, AMIPLANT GmbH, Germany) will be implanted into the capsular bag after removal of the of the natural lens. This IOL is CE-certified. Asphericity and dioptric power of the IOL are customized for each individual eye.

SUMMARY:
Cataract surgery in patients with irregular corneas presents unique challenges, primarily due to the high variability in keratometry and corneal tomography measurements, which complicates accurate intraocular lens (IOL) calculations. In these patients, therapeutic options are currently limited to either non-toric IOLs and rigid contact lenses postoperatively or conventional toric IOLs for the reduction of total astigmatism within cataract surgery. While conventional toric IOLs may be beneficial in selected cases with a stable astigmatic pattern and clear axis, their effectiveness is largely limited, as significant irregularity and higher order aberrations reduce predictability, accuracy of formulae, and refractive outcomes. Therefore, the development of a reliable method to reduce total astigmatism - including irregular components - would represent a major advancement, potentially improving both visual function and patient quality of life. The aim of this exploratory study is to evaluate the effectiveness of customized toric intraocular lenses (AMILens Individual, AMIPLANT GmbH, Germany) in reducing total corneal astigmatism in patients with a significant irregular astigmatic component. These lenses are designed to address corneal aberrations up to the 6th Zernike order, thereby extending correction beyond the capabilities of conventional toric IOLs. To our knowledge, no clinical study has yet investigated this novel approach.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Scheduled cataract surgery
* At least 1.75 D of total astigmatism in the CASIA2 measurement
* At least 0.75 D of asymmetry or higher order irregularity within the 6mm zone of the real (total) index corneal refractive map of the CASIA2 measurements

Exclusion Criteria:

* Relevant central corneal scars
* PEX, previous ocular surgery, severe trauma or any pathology that could lead to an unstable capsular bag
* Combined surgery (cataract plus glaucoma/vitreoretinal/corneal surgery)
* Postoperative best corrected distance visual acuity below 0.3 Snellen decimal
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change of Astigmatism | 4-8 weeks post-surgery
  The change of astigmatism is defined by the difference of the postoperative total refractive/ocular astigmatism (assessed via subjective refraction) to the preoperative corneal astigmatism (assessed via the utilized measurement devices).
  Reduction in total ocular (refractive) astigmatism will be quantified as both absolute reduction (Diopter) and relative reduction (%). Descriptive statistics will include mean, standard deviation, median, interquartile range, and range. Normality will be tested using the Shapiro-Wilk test and Q-Q plots.
  If normally distributed: comparisons between preoperative and postoperative values will be assessed with a paired t-test.
  If not normally distributed: the Wilcoxon signed-rank test will be applied. Results will be presented with 95% confidence intervals. As this is an exploratory study, p-values will be reported descriptively, and values below 0.05 will not be interpreted as statistically significant.

SECONDARY OUTCOMES:
Agreement of measured variables for astigmatism across devices | 4-8 weeks post cataract surgery
  The agreement of the variables anterior corneal astigmatism, posterior corneal astigmatism, total corneal astigmatism, Zernike Polynomials first to seventh order, lower order aberrations (LOAs), and higher order aberrations (HOAs) are compared across the utilized measurement devices Pentacam, Anterion, ms39, and CASIA2. All mentioned variables are on a ratio scale.
  Agreement between different devices will be assessed using: Bland-Altman analysis (mean difference and 95% limits of agreement),Intraclass correlation coefficients (ICCs) for reliability, and, where appropriate, repeated-measures ANOVA or Friedman test (non-parametric) across multiple modalities.
Change of higher order optical aberrations (HOAs) | 4-8 weeks post cataract surgery
  Higher order optical abberation values are measured posoperatively for the whole eye (cornea and lens) with the osiris device, and compared to the preoperative corneal higher order abberations, which are measured with the Casia2 and the ms39 devices.
  Reduction in higher order aberrations will be quantified as both absolute reduction (D) and relative reduction (%). The same descriptive statistics, normality testing, and comparison testing as described above will be applied. Results will be presented with 95% confidence intervals and p-values will be reported descriptively.
Surgically induced corneal astigmatism (SIA) | From enrollment to the end last study visit (4-8 weeks post surgery)
  Surgically induced corneal astigmatism (SIA) will be evaluated by calculating the vectorial changes of corneal astigmatism (magnitude ind diopter and axis in degree) between preoperative and postoperative corneal astigmatism measurements for each measurement device
Postoperative uncorrected and best-corrected distance visual acuity | 4-8 weeks post cataract surgery
  These values are assessed via standardized subjective refraction using the jackson cross cylinder method, and will be described descriptively in logMAR unit. Postoperative uncorrected and best-corrected visual acuity will be analyzed as both continuous variables and using threshold-based categories. Descriptive statistics will include mean, standard deviation, median, interquartile range, and range.

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Clinic, Department for Ophthalmology and Optometry, Linz, Austria

IPD SHARING:
Plan to Share IPD: No
The individual data will not be made available to other researchers. Only the results will be shared in peer-reviewed journals.